CLINICAL TRIAL: NCT03009591
Title: Prospective and Multicenter Study to Assess the Safety and Effectiveness of a Physiotherapy Treatment Through Fascial Therapy in Hemophilic Elbow Arthropathy. A Pilot Study.
Brief Title: Fascial Therapy in Elbow Hemophilic Arthropathy
Acronym: HeL-Fascial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Real Fundación Victoria Eugenia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HeL-Fascial
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hemophilia
Keywords: Hemophilia; Elbow; Arthropathy; Joint pain; Range of motion; Myofascial techniques; Safety patients; Quality of life; Functionality
MeSH Terms: conditions — Hemophilia A; Joint Diseases; Arthralgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expermiental group (Experimental): All patients included in the experimental group should be on prophylactic treatment with FVIII / FIX concentrates. Likewise, the factor should be administered on the same day that they receive each of the fascial therapy treatment sessions. Each session will last approximately 50 minutes, with three physiotherapy sessions taking place over a period of 3 weeks. The treatment program includes 11 maneuvers that must be administered bilaterally:
  Interventions: Other: Experimental group
- Control group (No Intervention): Subjects included in the control group will not receive physical therapy through fascial therapy and will continue with their usual routine of physical activity and exercise, and with the same pharmacological treatment regimen with FVIII / FIX. At the end of the study period the intervention will be applied under the same conditions as the experimental group, analyzing the overall sample at the end of the study.

INTERVENTIONS:
Other: Experimental group — Longitudinal surface sliding maneuver over the superficial fascia in the anterior region of the arm and the forearm. Applied in 3 strokes.
  * Transverse sliding of the flexor muscles of the wrist and fingers.
  * Transverse sliding for the biceps brachii muscle.
  * Longitudinal surface sliding over the superficial fascia in the posterior arm region.
  * Transverse sliding over the brachial triceps tendon.
  * Transverse sliding for the pectoralis major muscle.
  * Transverse sliding for the posterior axillary region pectoralis major muscle.
  * Induction of the posterior axillary fold.
  * Induction (crossed hands over the brachial region and forearm).
  * Maneuver of transverse planes for the cervicothoracic region.
  * Upper limb telescopic maneuver.
  Other Names: Fascial therapy group
  Arms: Expermiental group

SUMMARY:
Introduction: The common clinical manifestations of hemophilia are skeletal muscle bleeds, especially hematomas and hemarthrosis. Repeated episodes of joint bleeding in certain joints, causing a progressive joint deterioration. Secondary disorders to this joint degeneration include: biomechanical alterations, loss of range of movement and periarticular muscle atrophy.

Design. A prospective, multicenter and longitudinal pilot study to evaluate the efficacy of a treatment protocol with fascial therapy applied in patients with hemophilic arthropathy of the elbow.

Aimed: To evaluate the safety and efficacy of a physiotherapy treatment by fascial therapy in patients with hemophilic arthropathy of the elbow Patients: A total of 60 patients with hemophilia and prophylactic treatment will be recruited for inclusion in the study. Patients will be recruited in 6 centers, from different regions of Spain.

Intervention: Each session will last approximately 50 minutes, with three physiotherapy sessions taking place over a period of 3 weeks. The treatment program includes 11 maneuvers that must be administered bilaterally:

Measuring instruments and study variables: goniometric evaluation (range of movement); visual analog scale (joint pain); Haemophilia Joint Health Score (joint status); DASH Questionnaire (functionality of upper limbs); SF-36 Questionnaire (perception of quality of life). At the same time, the study will allow to determine joint bleeding caused by applied physiotherapy treatment.

Expected results: First, it is intended to demonstrate the safety of this physiotherapy technique in patients with hemophilia. Likewise, an improvement in the perception of elbow pain and joint mobility is expected. An improved functionality of the upper limb is also foreseen and with it, an enhanced perception of quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* Patients adults (over 18 years)
* Patients diagnosed with hemophilic arthropathy of the elbow (by clinical assessment with the Hemophilia Joint Health Score)
* Patients pn prophylactic treatment with FVIII / FIX concentrates.

Exclusion Criteria:

* Patients without ambulation ability
* Patients with inhibitors
* Patients with neurological or cognitive alterations that impede the comprehension of the questionnaires and physical tests
* Patients who have not signed the informed consent document.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline elbow joint bleeding frequency after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  After the first session of physiotherapy patients will be given a self-register where they can record all the observations they feel (from hematomas or hemarthros, to any other discomfort or perception). Similarly, the principal investigator of the study will monitor all patients within 48 hours after each physical therapy session.

SECONDARY OUTCOMES:
Change from baseline range of motion of elbow after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Change from range of movement of elbow during treatment and follow-up period at 3 months. The range of motion of the elbow joint will be measured using a universal goniometer, using the protocol for measuring joint motion described by Felipe Querol.
  Measurement instrument: universal goniometer with the protocol to measurement for patients with hemophilia
Change from baseline elbow joint status after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Change from elbow joint status during treatment and follow-up period at 3 months. Measurement instrument: Haemophilia Joint Health Score (scale 0-20).
Change from baseline joint pain of elbow after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Change from joint pain of ankle during treatment and follow-up period at 3 months.The perception of ankle pain will be measured using visual analog scale (scale 0-10).
Change from baseline upper limb functionality after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Change from upper limb functionality during treatment and follow-up period at 3 months. The perception of ankle pain will be measured using DASH Questionnaire. The Spanish version of this scale used internationally will evaluate upper limb functionality.
Change from baseline quality of life after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Change from quality of life during treatment and follow-up period at 3 months. The quality of life perception will be measured using SF-36 Questionnaire. This scale will assess the perception of quality of life of patients included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Eugenia Foundation, Madrid, Madird, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuesta-Barriuso R, Merono-Gallut J, Donoso-Ubeda E, Lopez-Pina JA, Perez-Llanes R. Effect of a Fascial Therapy Treatment on Quality of Life in Patients With Hemophilic Elbow Arthropathy: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 May;103(5):867-874. doi: 10.1016/j.apmr.2021.12.023. Epub 2022 Jan 23. PMID 35081366
- [Derived] Cuesta-Barriuso R, Perez-Llanes R, Lopez-Pina JA, Donoso-Ubeda E, Merono-Gallut J. Manual therapy reduces the frequency of clinical hemarthrosis and improves range of motion and perceived disability in patients with hemophilic elbow arthropathy. A randomized, single-blind, clinical trial. Disabil Rehabil. 2022 Jul;44(15):3938-3945. doi: 10.1080/09638288.2021.1894607. Epub 2021 Mar 8. PMID 33684015